CLINICAL TRIAL: NCT05217836
Title: Iron Metabolism Disorders in Patients With Sepsis or Septic Shock. Diagnosis and Monitoring of Treatment Based on Standard and New Laboratory Parameters.
Brief Title: Iron Metabolism Disorders in Patients With Sepsis or Septic Shock.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Czempik, Professor (assistant)/lecturer, Medical University of Silesia
Other Study IDs: PCN-2-083/N/O/K
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Anemia of Chronic Disease; Sepsis; Septic Shock
Keywords: ferritin; transferrin; transferrin saturation; hepcidin; reticulocyte hemoglobin content; parenteral iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Sepsis; Shock, Septic | interventions — Reticulocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ferritin; iron; transferrin; transferrin saturation; hemoglobin in reticulocyte; hepcidin — All patients will have the following laboratory parameters determined: ferritin, iron, transferrin, transferrin saturation, hemoglobin in reticulocyte, hepcidin. Patients with hemoglobin in reticulocyte below reference range will receive parenteral iron.

SUMMARY:
Anemia is a common health problem. Depending on a geographical region, anemia affects even 50% of population. Among patients admitted to the intensive care unit (ICU) anemia may affect as much as 66% of patients. Moreover, many patients develop anemia during the ICU stay. In general population the most common cause of anemia is iron deficiency (ID). The investigators lack information on the incidence of ID and anemia of inflammation (AI) with absolute ID (mixed type of anemia: AI + IDA) or functional ID (AI) in patients with sepsis or septic shock hospitalised in the ICU. Therefore, the aim of the study is to improve diagnosis of iron deficiency (ID) and anemia of inflammation (AI) with absolute ID (AI + IDA) or functional ID (AI) in patients with sepsis or septic shock.

ID have negative effects on the body and is associated with impaired production of proteins responsible for transport of oxygen in the blood (hemoglobin) and oxygen storage (myoglobin), and impaired immune function. Development of anemia is associated with well documented complications: organ hypoxia, myocardial infarction, stroke, infection. Replenishment of iron at this early stage may potentially prevent IDA. It is advantageous to replenish iron stores in order to avoid these complications, especially in patients with sepsis or septic shock. In IDA red blood cell transfusion is not recommended as it leads to other numerous complications. Therefore the patients presenting with laboratory results suggesting ID will receive divided doses od parenteral iron. Monitoring of iron replenishment will be based on a new laboratory parameter- reticulocyte hemoglobin equivalent.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sepsis or septic shock according to the third international definition and appropriate diagnostic criteria

Exclusion Criteria:

* active bleeding
* erythrocyte mean corpuscular volume (MCV) above the reference range
* diagnosed thalassemia or suspicion of thalassemia based on Mentzer index [9]
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the intensive care unit diagnosed with sepsis/septic shock
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess in patients with sepsis or septic shock the incidence of: iron deficiency, anemia of inflammation with absolute iron deficiency, anemia of inflammation with functional iron deficiency | Through study completion, an average of 1 year
  Incidence of the abovementioned conditions in numbers (%) in patients with sepsis or septic shock based on the results of hemoglobin, hepcidin, reticulocyte hemoglobin equivalent (RET-He)
To analyze associations between standard (ferritin; transferrin saturation) and new (hepcidin; reticulocyte hemoglobin equivalent) laboratory tests used in diagnosis of anemia in patients with sepsis or septic shock | Through study completion, an average of 1 year
  Presence or lack of correlation between the abovementioned laboratory tests
To assess the utility of a new diagnostic parameter of iron deficiency (reticulocyte hemoglobin equivalent) in monitoring treatment of iron deficiency in patients with sepsis or septic shock | Through study completion, an average of 1 year
  Assessment of the effect of divided doses of parenteral iron on concentration of reticulocyte hemoglobin equivalent (determinations performed in time intervals of 3-5 days) in patients with sepsis or septic shock
To assess the effect of divided doses of parenteral iron on anemia in patients with sepsis or septic shock without chronic kidney disease or acute kidney injury requiring renal replacement therapy | Through study completion, an average of 1 year
  Changes in hemoglobin concentration with consideration of iatrogenic blood loss (blood withdrew for laboratory tests)
To assess the effect of divided doses of parenteral iron and erythropoiesis- stimulating agent (epoetin alpha) on anemia in patients with sepsis or septic shock with chronic kidney disease or acute kidney injury requiring renal replacement therapy | Through study completion, an average of 1 year
  Changes in hemoglobin concentration with consideration of iatrogenic blood loss (blood withdrew for laboratory tests)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassebaum NJ, Jasrasaria R, Naghavi M, Wulf SK, Johns N, Lozano R, Regan M, Weatherall D, Chou DP, Eisele TP, Flaxman SR, Pullan RL, Brooker SJ, Murray CJ. A systematic analysis of global anemia burden from 1990 to 2010. Blood. 2014 Jan 30;123(5):615-24. doi: 10.1182/blood-2013-06-508325. Epub 2013 Dec 2. PMID 24297872
- [Background] Clark SF. Iron deficiency anemia. Nutr Clin Pract. 2008 Apr-May;23(2):128-41. doi: 10.1177/0884533608314536. PMID 18390780
- [Background] Corwin HL, Gettinger A, Pearl RG, Fink MP, Levy MM, Abraham E, MacIntyre NR, Shabot MM, Duh MS, Shapiro MJ. The CRIT Study: Anemia and blood transfusion in the critically ill--current clinical practice in the United States. Crit Care Med. 2004 Jan;32(1):39-52. doi: 10.1097/01.CCM.0000104112.34142.79. PMID 14707558
- [Background] Musallam KM, Taher AT. Iron deficiency beyond erythropoiesis: should we be concerned? Curr Med Res Opin. 2018 Jan;34(1):81-93. doi: 10.1080/03007995.2017.1394833. Epub 2017 Nov 3. PMID 29050512
- [Background] Czempik PF, Wojnarowicz O, Krzych LJ. Let us use physiologic transfusion triggers: Favorable outcome in an 86-year-old Jehovah's witness with a haemoglobin nadir of 44g L-1. Transfus Apher Sci. 2020 Apr;59(2):102718. doi: 10.1016/j.transci.2020.102718. Epub 2020 Jan 7. PMID 31926739
- [Background] Meybohm P, Richards T, Isbister J, Hofmann A, Shander A, Goodnough LT, Munoz M, Gombotz H, Weber CF, Choorapoikayil S, Spahn DR, Zacharowski K. Patient Blood Management Bundles to Facilitate Implementation. Transfus Med Rev. 2017 Jan;31(1):62-71. doi: 10.1016/j.tmrv.2016.05.012. Epub 2016 May 28. PMID 27317382
- [Background] Munoz M, Acheson AG, Auerbach M, Besser M, Habler O, Kehlet H, Liumbruno GM, Lasocki S, Meybohm P, Rao Baikady R, Richards T, Shander A, So-Osman C, Spahn DR, Klein AA. International consensus statement on the peri-operative management of anaemia and iron deficiency. Anaesthesia. 2017 Feb;72(2):233-247. doi: 10.1111/anae.13773. Epub 2016 Dec 20. PMID 27996086
- [Background] Wish JB. Assessing iron status: beyond serum ferritin and transferrin saturation. Clin J Am Soc Nephrol. 2006 Sep;1 Suppl 1:S4-8. doi: 10.2215/CJN.01490506. PMID 17699374
- [Background] Buttarello M. Laboratory diagnosis of anemia: are the old and new red cell parameters useful in classification and treatment, how? Int J Lab Hematol. 2016 May;38 Suppl 1:123-32. doi: 10.1111/ijlh.12500. Epub 2016 May 16. PMID 27195903
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Mentzer WC Jr. Differentiation of iron deficiency from thalassaemia trait. Lancet. 1973 Apr 21;1(7808):882. doi: 10.1016/s0140-6736(73)91446-3. No abstract available. PMID 4123424